CLINICAL TRIAL: NCT07230314
Title: Luminate Study: A Single-arm, Single-center, Open-label Clinical Study of Transarterial Chemoembolization (TACE) Plus Stereotactic Body Radiotherapy (SBRT) Combined With PD-1/L1 Inhibitor and Donafenib as First-line Therapy for Unresectable Hepatocellular Carcinoma.
Brief Title: Sequential Transarterial Chemoembolization (TACE), Stereotactic Body Radiation Therapy (SBRT), and Immune Checkpoint Inhibitors for Unresectable Hepatocellular Carcinoma Treated With Donafenib
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Liu Xiufeng, professor, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q81
Record Dates: First submitted 2025-09-29; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: transarterial chemoembolization (TACE); stereotactic body radiotherapy (SBRT); PD-1/L1 inhibitor; donafenib; first-line therapy
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE and SBRT combined with immune checkpoint inhibitors and treatment with donafenib (Experimental)
  Interventions: Drug: Donafina; Drug: PD-1/PD-L1 inhibitor

INTERVENTIONS:
Drug: Donafina — During the treatment, oral administration of Donafenib (0.2g, bid) was consistently administered
Drug: PD-1/PD-L1 inhibitor — According to the specific drug instructions, Q3W， The maximum usage time is 2 years

SUMMARY:
This study is a single arm, single center, open label clinical trial. Recruit 34 subjects who meet the inclusion criteria and receive hepatic artery chemoembolization (TACE) and stereotactic body radiotherapy (SBRT) combined with immune checkpoint inhibitors and donafenib treatment according to the study plan. The treatment cycle and dosage can be adjusted according to the patient's tolerance. Until disease progression or intolerable toxic reactions occur. Observe the effectiveness and safety indicators during the experimental process.

DETAILED DESCRIPTION:
This study is a single arm, single center, open label clinical trial. Recruit 34 subjects who meet the inclusion criteria and receive hepatic artery chemoembolization (TACE) and stereotactic body radiotherapy (SBRT) combined with immune checkpoint inhibitors and donafenib treatment according to the study plan. The treatment cycle and dosage can be adjusted according to the patient's tolerance. Until disease progression or intolerable toxic reactions occur. Observe the effectiveness and safety indicators during the experimental process.

Efficacy evaluation: The first efficacy evaluation is conducted 6 weeks (± 7 days) after the first administration, and every 6 weeks (± 7 days) thereafter. Imaging examinations include: CT or MRI of the brain, chest, abdomen (including pelvic cavity) (all are enhanced, unless contrast agents are contraindicated, plain scan can be used as a substitute).

Safety evaluation: Conducted on a weekly basis, objective indicators are obtained through examination, and subjective indicators are obtained through adverse events reported by patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 75 years old (including 18 and 75), with no gender restrictions;
2. Hepatocellular carcinoma diagnosed by histopathology, cytology or imaging;
3. Has not received any systemic anti-tumor therapy for the current stage of the disease in the past, including surgery (excluding stent placement), radiotherapy, chemotherapy, targeted therapy, immunotherapy, or investigational therapy;
4. CNLC staging Ib IIIa stage, cannot be surgically removed;
5. The maximum diameter of the tumor exceeds 5cm, and the number of tumors does not exceed 3 (1-3);
6. Can merge portal vein cancer thrombus;
7. Has not received any systemic anti-tumor therapy for the current stage of the disease in the past, including surgery (excluding stent placement), radiotherapy, chemotherapy, targeted therapy, immunotherapy, or investigational therapy;
8. Child Pugh score A5-B7;
9. ECOG (Eastern Cooperative Oncology Group) Physical Status Score: 0-1 points;
10. Expected survival period ≥ 3 months:
11. The main organ function is good, which meets the following criteria (no blood components, cell growth factors, white blood boosting drugs, platelet boosting drugs, or anemia correcting drugs are allowed to be used within 14 days before enrollment):

Neutrophils ≥ 1.5 × 109/L; White blood cell count ≥ 3.0 × 109/L; Platelets ≥ 100 × 109/L; Hemoglobin ≥ 90g/L; Serum albumin ≥ 34g/L; Total bilirubin ≤ 1.5 × ULN (for patients with biliary obstruction receiving biliary drainage, it can be relaxed to<2.5 × ULN); AST and ALT ≤ 2.5xULN (for patients with liver metastases, they can be relaxed to ≤ 5xULN); Creatinine clearance rate ≥ 60ml/min or blood creatinine ≤ 1.5 × ULN; INR ≤ 1.5 × ULN and APTT ≤ 1.5 × ULN (for stable dose anticoagulant therapy such as low molecular weight heparin or warfarin, and INR can be screened within the expected therapeutic range of anticoagulants); Electrocardiogram: QTc ≤ 450ms (male), ≤ 470ms (female); Cardiac ultrasound: LVEF (left ventricular ejection fraction) ≥ 50%; 8) Women of childbearing age must undergo a blood pregnancy test within 7 days before enrollment, and the result must be negative. They must also be willing to use appropriate contraception methods during the trial period and for 6 months after the end of treatment. For males, surgical sterilization should be performed, or they should agree to use appropriate contraception methods during the study period and within 3 months after the end of treatment; 9) Voluntarily participate in this study and sign an informed consent form; Good compliance, agree to cooperate and receive survival follow-up;

Exclusion Criteria:

1. Received any of the following treatments:

   Previously received ICIs and/or HDACi treatment; Received the last anti-cancer treatment (including surgery, radiation therapy, etc.) within 4 weeks before enrollment; Received any other experimental drug/device treatment within 4 weeks prior to enrollment; Simultaneously enrolled in another clinical study, unless it is an observational (non interventional) clinical study or an interventional clinical study follow-up;
2. Known patients who are allergic to the components of the investigational drug;
3. Patients known to have central nervous system metastases;
4. Severe gastrointestinal dysfunction (with bleeding, severe inflammation, obstruction, or diarrhea greater than grade 2);
5. Serious infections (CTC AE>grade 2) occurred within the first 4 weeks of enrollment, such as severe pneumonia, bacteremia, and infection complications that require hospitalization. Symptoms and signs of infection within the first 2 weeks of enrollment require intravenous antibiotic treatment (excluding prophylactic use of antibiotics);
6. Within the year prior to enrollment, there have been arterial/venous thrombotic events such as cerebrovascular accidents, deep vein thrombosis, and pulmonary embolism;
7. Clinical symptoms or diseases of the heart that have not been well controlled, such as: (1) NYHA grade 2 or above heart failure; (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within one year; (4) Patients with clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
8. Patients with malignant tumors other than liver cancer prior to the first use of the investigational drug are excluded, except for malignant tumors with low-risk metastasis and mortality risk (5-year survival rate>90%), such as fully treated cervical carcinoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma;
9. Merge active hepatitis B (HBV DNA ≥ 2000IU/mL or 104 copies/mL) and hepatitis C (positive for hepatitis C antibodies);
10. People who are known to have acquired immunodeficiency syndrome (AIDS) or HIV test positive, active syphilis infection;
11. Having a clear history of neurological or mental disorders, including epilepsy or dementia:
12. Planned pregnancy, pregnant and lactating women; According to the researchers' assessment, there may be other factors that could force the subjects to terminate the study midway, such as non-compliance with the protocol, having other serious illnesses (including mental illnesses) that require concomitant treatment, severe abnormal laboratory test values, family or social factors that may affect the safety of the subjects or the collection of trial data, etc;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, ORR | If the therapeutic effect reaches CR or PR, the subject must confirm it no less than 4 weeks ± 7 days after the initial evaluation.

SECONDARY OUTCOMES:
Overall survival, OS | every 3 months after the patient completed the trial treatment
disease control rate | If the therapeutic effect reaches CR or PR, the subject must confirm it no less than 4 weeks ± 7 days after the initial evaluation.